CLINICAL TRIAL: NCT03285282
Title: Evaluation of Thoracolumbar Interfascial Plane Block for Postoperative Analgesia After Herniated Lumbar Disc Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Lecture of anesthesia,intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 123/2017
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Analgesia After Disc Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Thoracolumber interfascial plane block
  Interventions: Procedure: Thoracolumber interfascial plane block
- Control (No Intervention)

INTERVENTIONS:
Procedure: Thoracolumber interfascial plane block — Thoracolumber interfascial plane block versus placebo
  Arms: Intervention

SUMMARY:
Several regional anesthesia have been shown to improve postoperative outcomes in many studies. The transversus abdominis plane (TAP) block provides anesthesia to the abdominal wall by introducing local anesthetic to the anterior rami of the spinal nerve roots. This work evaluates the analgesic effects gained after performing thoracolumbar interfacial plane block (analogous to the TAP block but intended for the back) which targets the sensory component of the dorsal rami of the thoracolumbar nerves in patients undergoing back surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA 1 or 2 aged between 21years old up to 60 years old of both sex scheduled of back surgery

Exclusion Criteria:

* Exclusion criteria will be patients refusal or inability to give an informed consent , history of relevant allergy to any of the drugs used in the procedure , previous lumbar spine surgery or back surgery with planed spinal fixation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | 24 hrs postoperative

SECONDARY OUTCOMES:
Total morphine consumption | 24 hrs postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided